CLINICAL TRIAL: NCT04663581
Title: Comparison Between the Right Lateral Decubitus and the Left Lateral Decubitus as Starting Position in Colonoscopy. Randomized Clinical Trial (POSCOL)
Brief Title: Comparison Between the Right Lateral Decubitus and the Left Lateral Decubitus as Starting Position in Colonoscopy
Acronym: POSCOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanitas University (Other)
Responsible Party: Principal Investigator, Claudia Aristizábal, Chief of Clinical Research Office, Sanitas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CEIFUS 597-19
Record Dates: First submitted 2020-12-03; First posted 2020-12-11 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Colonoscopy
Keywords: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Sided Colonoscopy (Experimental): Left Sided starting position in colonoscopy
  Interventions: Other: Left Sided Colonoscopy
- Right sided Colonoscopy (Active Comparator): Right Sided starting position in colonoscopy
  Interventions: Other: Right Sided Colonoscopy

INTERVENTIONS:
Other: Left Sided Colonoscopy — Starting colonoscopy with the patient in left decubitus
  Arms: Left Sided Colonoscopy
Other: Right Sided Colonoscopy — Starting colonoscopy with the patient in right decubitus
  Arms: Right sided Colonoscopy

SUMMARY:
Randomized Clinical trial between two positions to initiate colonoscopy, Right Sided vs Left Sided

DETAILED DESCRIPTION:
Objective To assess whether in the colonoscopy, the initial position of the patient in the right lateral decubitus (DLD) translates into advantages such as: shorter examination time or greater range of detection of polyps, compared to the left lateral decubitus (DLI), a position traditionally used.

Methodology This is a randomized and controlled clinical trial to be carried out in the city of Bogotá, in the Gastroenterology and Digestive Endoscopy Unit of the Colombia University Clinic, a fourth-level private clinic, a unit in which 7746 colonoscopies were performed in 2017.

The study will be carried out over a period of 2 months until the sample is completed.

Patients will be randomized to start their colonoscopy in the right lateral decubitus or left lateral decubitus and it would be assessed, the time to reach transverse colon, cecum and comfort perceived by the gastroenterologist and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for diagnostic colonoscopies in the digestive endoscopy unit.

Exclusion Criteria:

* Therapeutic colonoscopies.
* Patients with a history of colonic resection.
* Patients who cannot give their informed consent.
* Under 18 years old.
* Pregnant women.
* Patients with significant cardiopulmonary, renal or psychiatric disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Time to Reach Transverse Colon | During Procedure
  Time from starting of colonoscopy until endoscopist reaches transverse colon
Time to Reach Cecum | During Procedure
  Time from starting of colonoscopy until endoscopist reaches cecum

SECONDARY OUTCOMES:
Number of polyps | During Procedure
  Number of polyps detected in procedure
Number of diverticula | During Procedure
  Number of diverticula detected in procedure
Cecal Intubation | During Procedure
  Passage of the colonoscope tip to a point proximal to the ileocecal valve, so that the entire cecal caput, including the medial wall of the cecum between the ileocecal valve and appendiceal orifice, is visible
Endoscopist Comfort | During Procedure
  Comfort of the endoscopist measure in a 0 to 10 scale, being 0 not difficulty experienced, and 10 impossibility to intubate the appendix
Patient Comfort | During Procedure
  Comfort of the patient measure in a 0 to 10 scale, being 0 not discomfort experienced, and 10 unbearable discomfort experienced during procedure
Change position needed | During Procedure
  Necessity of changing starting position of the patient during procedure
Abdominal pressure needed | During Procedure
  Necessity of maneuvers to increasing abdominal pressure during procedure
Major adverse event | During Procedure
  Transient or Prolonged hypoxemia, Arrhythmias, Hypotension, Perforation.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universitaria Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided